CLINICAL TRIAL: NCT00204074
Title: Treatment of Menstrual Migraine With Sequential, Transdermal, 17-Beta-Estradiol. A Double-Blind, Randomised, Cross-Over Trial.
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Linkoeping (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Mensmig1
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2005-12-29 (Estimated); Status verified 2005-09

CONDITIONS: Migraine
Keywords: Migraine; Menstrual cycle; 17 beta-estradiol; Transdermal administration
MeSH Terms: conditions — Migraine Disorders | interventions — Estradiol; Pharmaceutical Preparations

INTERVENTIONS:
Drug: 17-beta-estradiol (drug)

SUMMARY:
The purpose of this study is to determine whether transdermally administered 17-beta estradiol sequentially could reduce the number of, and severity of, menstrual migraine attacks.

DETAILED DESCRIPTION:
During the fertile ages, migraine is more common in women than in men (3:1). Hormonal factors has been proposed to affect this difference and it has been shown that a rapid decrease in serum concentrations of estrogens might trigger an attack.About 15 percent of all women with migraine suffer from menstrual migraine which means that the attacks only come during the menstrual period and start +/- 24 hours of the bleeding start, i.e when there is a rapid decrease in serum concentrations of sex hormones.

Stabilizing the serum concentrations of estrogens seems to be crucial in the prophylactic treatment of menstrual migraine. A number of studies have focused on treatment with estradiol during the menstrual cycle but results are conflicting and doses and control groups have varied a lot. other studies have tried to reduce the exposition of estrogens by treatment with, for example, GnRH analogues. This treatment stabilizes the woman's serum concentrations of sex hormones on a very low level, like during the menopause, and it seems to be effective but there are a number of side-effects and the treatment is expensive.

Comparison: In a double-blind, randomized cross-over trial women with strictly defined menstrual migraine will receive treatment with 100 microg 17-beta estradiol/placebo transdermally one week before the estimated start of the menstrual bleeding and twoo weeks on. After three cycles and a wash-out period the treatment will be repeated but now with the tratment the woman did not have during the first treatment period. The women serve as their own controls.

ELIGIBILITY:
Inclusion Criteria:

* Migraine only during the menstrual period
* Migraine attacks each menstrual period during the last year
* Regular menstrual cycle

Exclusion Criteria:

* Migraine other times than during the menstrual period
* Use of hormonal contraceptives (other than depo-provera)during the last three months.
* Depo-provera injection the last year
* History of Thrombo-embolism
* Liver disease
* History of malignancy
* Breast-feeding during the last two months
* Abortion/miscarriage during the last two months
* Pregnancy

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Dates: Start 2001-10; Study Completion 2005-07

PRIMARY OUTCOMES:
Number of migraine attacks
Severeity of migraine attacks
Analgetics used

SECONDARY OUTCOMES:
Bleeding disturbances

CONTACTS AND LOCATIONS:
Overall Officials: Jan Brynhildsen, Principal Investigator — Department of Obstetrics & Gynecology, University Hospital, SE-58185, Linköping, Sweden
Locations (1):
- Division of Obstetrics & Gynecology, Department of Molecular and Clinical Medicine, Faculty of Health Sciences, Linköping, Sweden

REFERENCES:
- [Derived] Almen-Christensson A, Hammar M, Lindh-Astrand L, Landtblom AM, Brynhildsen J. Prevention of menstrual migraine with perimenstrual transdermal 17-beta-estradiol: a randomized, placebo-controlled, double-blind crossover study. Fertil Steril. 2011 Aug;96(2):498-500.e1. doi: 10.1016/j.fertnstert.2011.05.089. Epub 2011 Jun 24. PMID 21704313